CLINICAL TRIAL: NCT01540955
Title: Cognitive Rehabilitation Group Intervention for Breast Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-003446; JCCCID256 (Other: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2012-02-16; First posted 2012-02-29 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
Keywords: Reduce Cognitive Complaints; improve cognitive function; post-treatment breast cancer patients
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Intervention program (Experimental)
  Interventions: Behavioral: Improving Cognition with group intervention
- Wait-list control group (No Intervention): The wait-list-control group will also be able to participate in the group intervention, but not until after all the study visits have been completed.

INTERVENTIONS:
Behavioral: Improving Cognition with group intervention — Participants attend 5 weekly group sessions that are 2 hours each, delivered by a trained therapist. Sessions focus on specific aspects of attention, memory, multi-tasking and encoding. Homework assignments are practiced between classes. Goals are set for improved functioning.
  Arms: Group Intervention program

SUMMARY:
There are over 2 million breast cancer survivors in the US today. Along with extended survival, many women experience short and long-term after effects of treatment, which may decrease their quality of life and contribute to other health problems. Cognitive complaints---difficulties with memory, concentration, and planning-are commonly reported after adjuvant treatments for breast cancer. This study is designed to test the efficacy of a 5 week group-based cognitive rehabilitation intervention on improving cognitive complaints and test performance, in comparison to women who will receive the same intervention at a later time (wait-list control). Women will also have an EEG test performed before and after the intervention program to see if improvements in cognitive complaints and performance can be documented by examining the EEG.

DETAILED DESCRIPTION:
Previous pilot work (non-randomized, pre-post design) has shown that this intervention was effective in improving post-intervention cognitive complaints and neuropsychological (NP) test performance. Because practice effects may influence NP performance, it is important to compare the intervention participants to women who are not exposed to the intervention. Thus, this randomized controlled trial will compare the active intervention to a control group of patients who will receive the intervention at a delayed time point. The primary outcomes are improvements in cognitive complaints and NP test performance 2 months after completion of the intervention program. Quantitative EEG (QEEG) measurements will be used as a secondary exploratory endpoint to see if this may be an effective biomarker of cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* age 21-65 years
* stage I, II, III breast cancer diagnosis within the past 18 months to 5 years
* currently disease free, but may be on endocrine therapy
* with evidence of need of cognitive therapeutic intervention, as demonstrated by mild or greater cognitive deficiencies on an objective screening measure
* reads and writes English
* able to give informed consent
* willing and able to attend 5 weekly group sessions and participate in pre and post-evaluation that will take place on the UCLA campus

Exclusion Criteria:

* evidence of uncontrolled depression

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cognitive function measured by neuropsychological assessment 2 months after group intervention | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Ganz, M.D., Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA, Los Angeles, California, United States